CLINICAL TRIAL: NCT03842982
Title: Phase III Randomized Clinical Trial Evaluating Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Ovarian Cancer Considering Two Different Settings: Primary Debulking Surgery (PDS) and Interval Debulking Surgery (IDS)
Brief Title: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Ovarian Cancer (CHIPPI)
Acronym: CHIPPI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIPPI-1808; 2018-003680-62 (EudraCT Number)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Ovary Neoplasms; Ovarian Cancer; Ovarian Carcinoma
Keywords: Ovarian cancer; Hyperthermic intraperitoneal chemotherapy; HIPEC; Primary Debulking Surgery; Interval Debulking Surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (PDS or IDS + HIPEC) (Experimental): Surgery (Primary Debulking Surgery (PDS) or Interval Debulking Surgery (IDS)) + Neo or Adjuvant chemotherapy (standard care) + HIPEC (hyperthermic intraperitoneal chemotherapy)
  Patients in this experimental arm will receive surgery (either PDS or IDS) and Neo and/or Adjuvant chemotherapy (CT) (as per standard care) combined with HIPEC. Patients undergoing PDS will also be receiving 6 cycles adjuvant CT according to the standard care (ideally 6 weeks post-surgery).
  Patient undergoing IDS will start with 6 cycles of neo-adjuvant CT with a 3 - 5 weeks washout period (4 - 6 weeks if administered Bevacizumab) prior to surgery. They may also undergo additional adjuvant CT post-surgery according to the standard care.
  Interventions: Drug: HIPEC
- Arm B (PDS or IDS) (No Intervention): Surgery (Primary Debulking Surgery (PDS) or Interval Debulking Surgery (IDS)) + Neo or Adjuvant chemotherapy ONLY (standard care, without HIPEC)
  Patients in the control group will ONLY receive the standard care, which consists of surgery (PDS or IDS) with Neo and/or Adjuvant chemotherapy (CT). Patients undergoing PDS will be receiving 6 cycles adjuvant CT according to the standard care (ideally 6 weeks post-surgery).
  Patient undergoing IDS will start with 6 cycles of neo-adjuvant CT with a 3 - 5 weeks washout period (4 - 6 weeks if administered Bevacizumab) prior to surgery. They may also undergo additional adjuvant CT post-surgery according to the standard care.

INTERVENTIONS:
Drug: HIPEC — HIPEC protocol (ONLY Arm A) consisted in cisplatin 100mg/m2 intraperitoneally (IP), heated to 40°C for 90 minutes, along with an IV perfusion of sodium thiosulfate.
  Administration of the dose should be according the following schedule:
  * 50% of the dose at start of perfusion, 25% of the dose after 30 minutes from start of the perfusion and 25% of the dose after 60 minutes from start of the perfusion.
  * The procedure takes 120 minutes with a 90-minute perfusion period. The IV perfusion of sodium thiosulfate is for renal protection. At the start of HIPEC procedure, 9 g/m2 in 200 ml of distilled water will be administered by IV over 15 to 30 minutes. It will be then followed by 12 g/m2 in 1 liter (1L) distilled water in a continuous IV for 6 hours.
  Other Names: Hyperthermic intraperitoneal chemotherapy
  Arms: Arm A (PDS or IDS + HIPEC)

SUMMARY:
This is a phase III, multicenter, interventional and randomized study which evaluates the use of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) coupled with either Primary Debulking Surgery (PDS) or Interval Debulking Surgery (IDS), in patients with ovarian cancer. This study aims to assess the efficacy, in terms of disease-free survival (DFS), the use of HIPEC combined with standard care (PDS or IDS) or standard care alone.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy, in terms of disease-free survival (DFS), the use of HIPEC treatment combined with standard care (PDS or IDS) or standard care alone (PDS or IDS alone).

Secondary objectives of the study include:

* Evaluating the efficacy of HIPEC in terms of overall survival (OS) in combination with standard of care
* Evaluating the morbidity associated with HIPEC.
* Evaluating the trade-off between efficacy and morbidity using the Q-TWiST approach.
* Evaluating the impact of HIPEC in terms of quality of life.

Exploratory objectives (optional) include:

* Evaluating the impact of HIPEC on the count of residual viable cells (evaluated by flow cytometry) in abdominal drainage fluids for patients recruited in Centre Oscar Lambret only.
* Constituting a biobank (tumoral samples and blood samples) for future translational researches

ELIGIBILITY:
Inclusion Criteria:

Pre-eligibility criteria to be checked before surgery for pre-registration

1. Age ≥18 years and ≤ 76 years
2. Histologically proven primary epithelial ovarian carcinoma or fallopian tube carcinoma or peritoneal carcinoma (including serous papillary adenocarcinoma, clear-cell carcinoma, mucinous adenocarcinoma and endometrioid carcinoma)
3. Pre-therapeutic FIGO (International Federation of Gynecology and Obstetrics) stage III
4. Patient eligible for

   1. Primary Debulking Surgery (PDS) with planned adjuvant chemotherapy +/- bevacizumab or other targeted therapy
   2. Or Interval Debulking Surgery (IDS) after neo-adjuvant chemotherapy +/- bevacizumab or other targeted therapy, with or without planned adjuvant chemotherapy +/- bevacizumab or other targeted therapy. In case of neo-adjuvant chemotherapy, surgery should be performed in a time interval of 3 to 5 weeks in case of chemotherapy without bevacizumab, and in a time interval of 4 to 6 weeks if chemotherapy is combined with bevacizumab. The patient remains eligible for the study if surgery is delayed beyond the recommended time interval.
5. WHO (World Health Organization Performance Status) ≤ 2
6. Physical status score ASA (American Society of Anesthesiologists) ≤ 2
7. Adequate bone marrow and renal function, as evidenced by the following tests performed within 7 days prior to surgery:

   * Absolute Neutrophil Count (ANC) ≥1,500/mm3
   * Platelets ≥100,000/mm3
   * Aspartate aminotransferase (ALT)/ Alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN) (≤5.0 × ULN in case of liver metastases)
   * Total bilirubin ≤1.5 × ULN (except in case of Gilbert's disease)
   * Creatinine clearance ≥ 60 mL/ min
8. Negative serum pregnancy test within 7 days prior to surgery for women of childbearing potential. For non-menopausal women, if no hysterectomy is planned, willing to accept the use of an effective contraceptive regimen during the treatment period and at least 6 months after the end of treatment (surgery or adjuvant chemotherapy)
9. Absence of contraindication to receive the products used in this study (cisplatin and products used in neo-adjuvant/ adjuvant chemotherapy) according to the most recent SmPC (Summary of Product Characteristics) of these products
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up
11. Signed written informed consent
12. Patient covered by the French or Belgian "Social Security" regime Criteria to be checked per-operatively for confirmation of enrolment and randomization
13. Residual disease after surgery (cytoreduction score CC) CC-0 (no macroscopic residue) or CC-1 (residue < 2.5 mm)
14. Per-operative hemorrhage < 2.5 L
15. Strictly less than 3 digestive resections performed during surgery
16. Diuresis maintained during surgery, without oliguria or anuria (per-operatory diuresis ≥ 0,5 mL/ kg/ h)

Exclusion Criteria:

1. Benign disease, borderline disease, non epithelial ovarian carcinoma or carcinosarcoma
2. Cirrhosis
3. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
4. Auditory impairment
5. Dehydration or intercurrent disease that contraindicates hyperhydration (including cardio-respiratory disease)
6. Other uncontrolled intercurrent disease including, but not limited to: diabetes; hypertension; symptomatic congestive heart or pulmonary failure; renal, hepatic or severe gastrointestinal (associated with diarrhea) chronic disease
7. Any unresolved NCI-CTCAE Grade ≥ 2 toxicity from previous anticancer therapy (excluding alopecia)
8. Concomitant treatment with prophylactic phenytoin
9. Receipt of live attenuated vaccine, including yellow fever vaccine, within 30 days prior to inclusion (and, if patient is enrolled, up to 30 days after the last administration of study treatment)
10. Pregnant or breastfeeding woman
11. Psychiatric illness or social situation that would limit compliance with study requirement, substantially increase the risk of side effects, or compromise the ability of the patient to give written informed consent
12. Inability to comply with medical follow-up of the trial (geographical, social or psychic reasons)
13. Person under guardianship

Ages: 18 Years to 76 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with ovarian cancer
Enrollment: 362 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | From randomization to first progression, relapse or death from any cause, whichever came first, assessed up to 5 years. (Follow-up up to 5 years)
  The DFS will be measured to assess the efficacy of the combination treatment of surgery and HIPEC or standard care alone.

SECONDARY OUTCOMES:
Overall survival | From randomization to first progression, relapse or death from any cause , whichever came first, assessed up to 5 years..
  The overall survival will be measured to assess the efficacy of HIPEC in combination with standard care.
Adverse events (AE) | Covers the whole treatment duration from Randomization up to the end of treatment (surgery or CT) plus 30 days.
  The adverse events (AE) are collected to evaluate the impact of HIPEC on the safety and on the feasibility of adjuvant treatment (if any) is planned after surgery.
Q-TWiST | Over the 5 year surveillance period
  Q-Twist (Quality-adjusted time without symptoms of disease or toxicity) will be calculated from the survival tile (OS and DFS) and AE (adverse events) data.
Quality of life of the patient (QLQC30) | Up to 2 years after the end of treatment (every 3 month)
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Score 30 (QLQ-C30) will be used to measure the quality of life of the patients.
Quality of life of the patient (QLQOV28) | Up to 2 years after the end of treatment (every 3 month)
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Ovarian Cancer Module (QLQ-OV28) will be used to measure the quality of life of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice NARDUCCI, MD, Study Director — Centre Oscar Lambret, Lille, France
Locations (18):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires St-Luc, Institut Roi Albert II, Brussels
- France (16):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Hôpital Jeanne de Flandre, Lille
  - Institut Paoli Calmettes, Marseille
  - ICM-Val d'Aurelle, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Clinique Mathilde, Rouen
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Hôpital de Hautepierre, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No